CLINICAL TRIAL: NCT00466206
Title: Phase II Magnetic Alteration of Pectus Excavatum
Brief Title: Magnetic Mini-Mover Procedure to Treat Pectus Excavatum
Acronym: 3MP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Harrison, Professor of Surgery and Pediatrics, Emeritus, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD 003341
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Pectus Excavatum
Keywords: pectus excavatum; magnetic alteration; chest wall deformity
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3MP - Treatment Arm (Experimental): Magnetic Mini-Mover Procedure using the Magnimplant and Magnatract
  Interventions: Device: Magnetic Mini-Mover Procedure (3MP); Device: Magnatract (external magnet in a removable external brace); Procedure: 3MP (Magnetic Mini-Mover Procedure)

INTERVENTIONS:
Device: Magnetic Mini-Mover Procedure (3MP) — A rare earth magnet encased in FDA-approved titanium will be implanted securely on the outer surface of the lower end of the sternum in patients with pectus excavatum. This is accomplished as an outpatient procedure, under brief general anesthesia.
  A 2-inch transverse skinline incision is made at the junction of the sternum and xyphoid and the space in front and behind the sternum is dissected bluntly. The titanium can containing the magnet is securely fixed to the sternum by screwing it into a titanium fixation disk in front of the sternum. The procedure takes 1/2-hour, and the patient can go home the same day.
  In another outpatient procedure, the Magnimplant is explanted 18 months after implantation.
  Other Names: 3MP
Device: Magnatract (external magnet in a removable external brace) — An external orthotic device "Magnatract" which includes an external magnet in a removable brace is fitted specifically to the patient's chest wall deformity. A calibrated meter in the external device measures the force applied between the two magnets. When the patient and family are comfortable with the device and comfort and skin condition have been assessed, the patient will be allowed to take the Magnatract home and begin the process of gradually advancing the sternum forward as the abnormal costal cartilage is reformed.
  Other Names: Magnetic Mini-mover
Procedure: 3MP (Magnetic Mini-Mover Procedure) — * Subject has EKG performed to measure baseline cardiac activity.
  * Magnimplant is implanted.
  * After one week, "Magnatract" is fitted.
  * Chest x-ray and 2nd EKG performed 30 days post-implantation.
  * Patient and parents complete QoL questionnaire 30d post-implantation.
  * Patient seen weekly for first month post-implantation to assess comfort and skin condition. Thereafter, will be seen monthly.
  * At each monthly visit, patient will have lateral and anterior-posterior chest X-rays to monitor sternal correction.
  * At each visit data logger is downloaded to measure strength of pull since last visit and amount of wear-time.
  * Magnimplant explanted 18 months later as 1/2-hr outpatient procedure.
  * CT scan and third EKG performed after explanation.
  * Patient and parents complete QOL questionnaires after explantation and 1 yr post-explantation.
  Other Names: 3MP

SUMMARY:
This is a medical research study.

The study investigators have developed a method to gradually repair pectus excavatum (sunken chest) deformity by placing a magnet on the sternum (breastbone) and then applying an external magnetic force that will pull the sternum outward gradually.

Potential candidates for this study are children and adolescents with a previously diagnosed congenital pectus excavatum (sunken chest) deformity who are otherwise healthy and are seeking corrective surgery for their condition. They will be residents of the U.S. and between the ages of 8 and 14 years of age. Potential candidates and their families will have already been counseled about this condition and about the standard way to repair this deformity.

The purpose of this study is to test what effects, good and/or bad, placing an external/internal magnetic device has on correcting pectus excavatum deformity in children, and the safety of using such a device for treatment.

DETAILED DESCRIPTION:
Pectus excavatum is the most common congenital chest wall abnormality in children. Surgical correction requires a big operation under general anesthesia which forces the sternum forward and holds it in place using a metal chest wall strut. Deformation of the chest wall under great pressure may result in complications and potential relapses as well as postoperative pain requiring hospitalization for regional and narcotic anesthesia for up to a week. An alternative principle for correction of chest wall and other deformities is gradual (bit-by-bit) correction using minimal force applied over many months (like moving teeth with orthodontic braces).

The hypothesis of this study is that constant outward force on the deformed cartilage in pectus excavatum will produce biologic reformation of cartilage and correction of the chest wall deformity.

The study investigators have developed a novel method of achieving gradual deformation/reformation of chest wall cartilage without the need for transdermal orthopedic devices or repeated surgeries. A magnetic force field is used to apply controlled, sustained force to promote biologic reformation of structural cartilage (the same principle as distraction osteogenesis). A magnet is implanted on the sternum and secured using a novel fixation strategy that can be accomplished through a 3-cm subxyphoid incision as a brief outpatient procedure. The magnet (and sternum) is pulled outward by another magnet suspended in a novel, low-profile, lightweight device previously molded to the patient's anterior chest wall. The external magnet allows individual adjustment in small increments of the distance (and, thus, force) and orientation of the force applied to the sternum. The low-profile, non-obtrusive anterior chest wall prosthesis is held in place by the force field between the two magnets.

The study objectives are to test the safety and probable benefit of this procedure in 10 otherwise healthy, young patients, between 8 years and 14 years of age, who have chosen to have this deformity corrected using this novel technique rather than the standard Ravitch or Nuss techniques. We will document the rate of correction by chest imaging and measurement of the Pectus Severity Index. The study investigators will document safety and efficacy with an EKG prior to implantation, one month post-implantation, and finally after the magnet is removed, as well as patient and family satisfaction with a post-procedure Quality of Life-type survey.

ELIGIBILITY:
Residents of the United States with previously diagnosed pectus excavatum who are referred to the UCSF Pediatric Surgery Service for evaluation and treatment will be considered for participation in this study. Only patients with moderate to severe pectus excavatum who meet all the inclusion criteria will participate. The patient and family will be fully counseled and consented about the risks and benefits of participation in the study, and will be asked to sign an informed consent reviewed and approved by the UCSF Committee on Human Research.

Inclusion Criteria:

1. Resident of the U.S.;
2. Otherwise healthy male or female with pectus excavatum deformity;
3. Between 8 and 14 years of age;
4. Pectus Severity Index > 3.5 (normal 2.56); and
5. Ability to read and speak English.

Exclusion Criteria:

1. Other congenital anomalies (including significant skeletal anomalies such as scoliosis, bony fusion involving the cervical vertebrae) not directly related to pectus excavatum;
2. Bleeding disorders;
3. Heart disease (including arrhythmia);
4. Persons with active implantable medical devices (AIMD) such as pacemakers;
5. Persons with a relative(s) or close family friend(s) living within their households and having a pacemaker;
6. Persons with arteriovenous malformations;
7. Chest deformity more complicated than pectus excavatum (e.g.. Poland syndrome);
8. Persons for whom a foreign body implant would pose a risk (e.g., immunodeficiency);
9. Persons at increased risk for general anesthesia (e.g., history of malignant hyperthermia);
10. Respiratory conditions that have required steroid treatment (e.g., prednisone)in the last 3 years;
11. Pregnancy;
12. Inability to understand or follow instructions;
13. Refusal to wear the external brace;
14. Inability to obtain pre-approval (authorization) from the patient's insurance carrier; and
15. Inability or refusal to return to UCSF for weekly follow-up visits for the first month after surgery.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2010-05 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Harrison, MD, Principal Investigator — University of California, San Francisco Medical Center and Children's Hospital
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] RAVITCH MM. The operative treatment of pectus excavatum. J Pediatr. 1956 Apr;48(4):465-72. doi: 10.1016/s0022-3476(56)80075-9. No abstract available. PMID 13295996
- [Background] WELCH KJ. Satisfactory surgical correction of pectus excavatum deformity in childhood; a limited opportunity. J Thorac Surg. 1958 Nov;36(5):697-713. No abstract available. PMID 13588724
- [Background] Morshuis WJ, Mulder H, Wapperom G, Folgering HT, Assman M, Cox AL, van Lier HJ, Vincent JG, Lacquet LK. Pectus excavatum. A clinical study with long-term postoperative follow-up. Eur J Cardiothorac Surg. 1992;6(6):318-28; discussion 328-9. doi: 10.1016/1010-7940(92)90149-r. PMID 1616728
- [Background] ADKINS PC, BLADES B. A stainless steel strut for correction of pectus escavatum. Surg Gynecol Obstet. 1961 Jul;113:111-3. No abstract available. PMID 13681493
- [Background] Shamberger RC. Congenital chest wall deformities. Curr Probl Surg. 1996 Jun;33(6):469-542. doi: 10.1016/s0011-3840(96)80005-0. No abstract available. PMID 8641129
- [Background] Nuss D, Croitoru DP, Kelly RE Jr, Goretsky MJ, Nuss KJ, Gustin TS. Review and discussion of the complications of minimally invasive pectus excavatum repair. Eur J Pediatr Surg. 2002 Aug;12(4):230-4. doi: 10.1055/s-2002-34485. PMID 12368998
- [Background] Beiser GD, Epstein SE, Stampfer M, Goldstein RE, Noland SP, Levitsky S. Impairment of cardiac function in patients with pectus excavatum, with improvement after operative correction. N Engl J Med. 1972 Aug 10;287(6):267-72. doi: 10.1056/NEJM197208102870602. No abstract available. PMID 5038952
- [Background] Lawson ML, Cash TF, Akers R, Vasser E, Burke B, Tabangin M, Welch C, Croitoru DP, Goretsky MJ, Nuss D, Kelly RE Jr. A pilot study of the impact of surgical repair on disease-specific quality of life among patients with pectus excavatum. J Pediatr Surg. 2003 Jun;38(6):916-8. doi: 10.1016/s0022-3468(03)00123-4. PMID 12778393
- [Background] Wynn SR, Driscoll DJ, Ostrom NK, Staats BA, O'Connell EJ, Mottram CD, Telander RL. Exercise cardiorespiratory function in adolescents with pectus excavatum. Observations before and after operation. J Thorac Cardiovasc Surg. 1990 Jan;99(1):41-7. PMID 2294364
- [Background] Haller JA Jr, Loughlin GM. Cardiorespiratory function is significantly improved following corrective surgery for severe pectus excavatum. Proposed treatment guidelines. J Cardiovasc Surg (Torino). 2000 Feb;41(1):125-30. PMID 10836238
- [Background] Zhao L, Feinberg MS, Gaides M, Ben-Dov I. Why is exercise capacity reduced in subjects with pectus excavatum? J Pediatr. 2000 Feb;136(2):163-7. doi: 10.1016/s0022-3476(00)70096-5. PMID 10657820
- [Background] Mead J, Sly P, Le Souef P, Hibbert M, Phelan P. Rib cage mobility in pectus excavatum. Am Rev Respir Dis. 1985 Dec;132(6):1223-8. doi: 10.1164/arrd.1985.132.6.1223. PMID 4073662
- [Background] Shamberger RC. Cardiopulmonary effects of anterior chest wall deformities. Chest Surg Clin N Am. 2000 May;10(2):245-52, v-vi. PMID 10803331
- [Background] Malek MH, Fonkalsrud EW, Cooper CB. Ventilatory and cardiovascular responses to exercise in patients with pectus excavatum. Chest. 2003 Sep;124(3):870-82. doi: 10.1378/chest.124.3.870. PMID 12970011
- [Background] Hebra A, Swoveland B, Egbert M, Tagge EP, Georgeson K, Othersen HB Jr, Nuss D. Outcome analysis of minimally invasive repair of pectus excavatum: review of 251 cases. J Pediatr Surg. 2000 Feb;35(2):252-7; discussion 257-8. doi: 10.1016/s0022-3468(00)90019-8. PMID 10693675
- [Background] Park HJ, Lee SY, Lee CS. Complications associated with the Nuss procedure: analysis of risk factors and suggested measures for prevention of complications. J Pediatr Surg. 2004 Mar;39(3):391-5; discussion 391-5. doi: 10.1016/j.jpedsurg.2003.11.012. PMID 15017558
- [Background] Weber TR. Further experience with the operative management of asphyxiating thoracic dystrophy after pectus repair. J Pediatr Surg. 2005 Jan;40(1):170-3. doi: 10.1016/j.jpedsurg.2004.09.039. PMID 15868580
- [Background] Fonkalsrud EW, Reemtsen B. Force required to elevate the sternum of pectus excavatum patients. J Am Coll Surg. 2002 Oct;195(4):575-7. doi: 10.1016/s1072-7515(02)01245-0. No abstract available. PMID 12375767
- [Result] Kowalewski J, Barcikowski S, Brocki M. Cardiorespiratory function before and after operation for pectus excavatum: medium-term results. Eur J Cardiothorac Surg. 1998 Mar;13(3):275-9. doi: 10.1016/s1010-7940(97)00326-6. PMID 9628377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Physician- or self-referral to the Chest Wall Deformity Clinic at UCSF for evaluation of pectus excavatum. Active recruitment from 2007-2009 to accrue ten subjects.
Groups:
- 3MP Treatment Arm: Undergo active Magnetic Mini-Mover Procedure for treatment of pectus excavatum. Active treatment = 18 months
Period: Overall Study
Arm/Group | 3MP Treatment Arm
Started | 10
Completed | 10 (One of 10 patients withdrawn from study but completed treatment under Compassionate Use Designation)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3MP Treatment Arm
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants] — Between 8 and 14 years of age
  Participants
    <=18 years | 10
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Affect on Cardiac Activity
Description: EKG performed prior to implantation, one month post-implantation, and after explanation to evaluate whether magnetic field near the heart adversely affects cardiac activity. Outcome measure describes number of patients who experienced adverse change in EKG.
Time Frame: One month post-explantation
Population: Per protocol, this is a single-arm, pilot study of ten subjects.
Measure: Number; unit: participants
Groups:
- Magnetic Mini-Mover Group: Treatment for pectus excavatum using Magnimplant and Magnatract
Arm/Group | Magnetic Mini-Mover Group
Number analyzed (Participants) | 10
participants | 0

2. Secondary Outcome: Patient Compliance
Description: Compliance measured by average number of hours per day external device was worn by patient, as measured by the data sensor and logging device built into external prosthetic
Time Frame: 18 months active Rx
Population: Per protocol
Measure: Mean (Full Range); unit: avg hours per day brace worn
Groups:
- Treatment Arm: Magnetic Mini-Mover Procedure
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
avg hours per day brace worn | 16 [11 to 23]

3. Primary Outcome: Damage/Discoloration to Skin
Description: Outcome measure is number of patients who experienced permanent skin damage or discoloration due to external brace wear
Time Frame: One-month post-explant
Population: Per protocol
Measure: Number; unit: participants
Groups:
- 3MP Treatment Group: Treatment of pectus excavatum with the Magnetic Mini-Mover Procedure
Arm/Group | 3MP Treatment Group
Number analyzed (Participants) | 10
participants | 0

4. Primary Outcome: Efficacy: Patient Satisfaction
Description: Based on patient response to one-year post-explantation QoL questionnaire: How satisfied are you with the correction of your chest? Ratings: 5-very satisfied; 4-satisfied; 3-unsure; 2-dissatisfied; 1-very dissatisfied
Time Frame: One year post-explant
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- 3MP Treatment Arm: Pectus excavatum treated with Magnetic Mini-Mover Procedure. Active treatment = 18 months
Arm/Group | 3MP Treatment Arm
Number analyzed (Participants) | 10
Scores on a scale | 3.7 (1.1)

5. Primary Outcome: Efficacy: Patient Recommendation of Treatment
Description: Based on patient response to one-year post-explantation QoL statement: "I would recommend this treatment for pectus excavatum (sunken chest) to someone else with pectus excavatum." Ratings: 5-strongly agree; 4-agree; 3-unsure; 2-disagree; 1-strongly disagree
Time Frame: One year post-explanation
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Magnetic Mini-Mover Group
Number analyzed (Participants) | 10
Scores on a scale | 4.2 (0.8)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Magnetic Mini-Mover Treatment: Use of the Magnimplant and Magnatract to treat pectus excavatum
Arm/Group | Magnetic Mini-Mover Treatment
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnetic Mini-Mover Treatment (N=10)
Wound infection (Surgical and medical procedures) | 3 (3)
Re-operation (Surgical and medical procedures) | 5 (6) — Re-operation to loosen overtightened implant; reattach or replace non-functional device; removal of devices that had a mechanical failure

LIMITATIONS AND CAVEATS:
Technical problems with measurement of PSI. PSI is uninformative in assessing efficacy of treatment as it is a dynamic measure that varies with patient position and respiration at any given measurement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No